CLINICAL TRIAL: NCT06507358
Title: Exploring the Sensory Experiences and Enhancement of Parent-Child Interaction in Garding Activities for Early Intervention in Preschool Children
Brief Title: Parent-Child Interaction in Garding Activities for Early Intervention Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N202405063
Record Dates: First submitted 2024-07-10; First posted 2024-07-18 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-05

CONDITIONS: Development Delay
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Intervention Model Description: A sampling will assign participants equally to a gardening group (Parent-Child Interaction) (N=30) and a waiting group (N=30). The gardening group (Parent-Child Interaction) will participate in group gardening activities for six to eight weeks, while the waiting group will join after eight-weeks waiting period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parent-Child Interaction group (Experimental): Inclusion criteria for the experimental group are as follows: (1) Children currently undergoing early intervention; (2) Children experiencing sensory processing issues and caregivers (including grandparents and great-grandparents) seeking to establish parent-child relationships or enhance self-efficacy; (3) Ability to participate on duration of interventive class and to comply with trial procedures and complete home assignments, having attended at least 3/4 of the sessions.
  Interventions: Behavioral: Parent-Child Interaction group
- Control group (No Intervention): Exclusion criteria for study participants are as follows: (1) Children aged under 4 or over 7 years; (2) Caregivers (including grandparents and great-grandparents) unable to communicate or read in Chinese. (3) Inability to participate on duration of interventive class.

INTERVENTIONS:
Behavioral: Parent-Child Interaction group — The intervention for the Parent-Child Interaction group consists of a 6-week program involving weekly 40-minute sessions of therapeutic horticulture in a group setting, with 4-6 participants per group. The sessions focus on sensory-motor activities aimed at helping children engage in daily tasks and activities. Various sensory stimuli are provided through different materials used in gardening activities, including visual, auditory, gustatory, tactile, and olfactory stimuli. The program encourages mutual support and sharing among group members, showcases different outcomes, and emphasizes a sense of responsibility for home care. With a family-centered approach, parental involvement serves as a mediator to promote children's overall development and abilities. Participants are required to complete homework assignments and maintain activity records, including documentation of the 6 sessions through photos and written records.
  Arms: Parent-Child Interaction group

SUMMARY:
Post-COVID-19, children's reduced interaction with nature has hindered their sensory development, particularly affecting those with developmental delays. This creates challenges for caregivers and impacts the children's abilities and parental mental health. While caregiver-centered interventions are known to benefit child development and reduce parent stress, there is a lack of such multidisciplinary programs in early intervention practices. This project investigates the impact of gardening activities on caregiver stress, self-efficacy, relationships, and parent-child conflict. Caregivers of children in early intervention in northern outpatient clinics will be recruited and randomly assigned to a gardening group or a waiting group. The gardening group will participate in activities for six to eight weeks, with assessments conducted before and after the intervention using various scales. Data will be analyzed using SPSS (Version 20.0) with a 0.05 significance level. Results will be shown as mean ± standard deviation. Descriptive statistics will analyze basic data and assessment items. The Chi-square test, Mann-Whitney U test, and Kruskal-Wallis ANOVA will compare outcomes. Spearman's rank correlation will assess relationships between caregivers' and children's data, caregiver efficacy, stress, and children's sensory interaction.

DETAILED DESCRIPTION:
Background:Following the COVID-19 pandemic, children have had significantly reduced interactions with nature, leading to a lack of sensory experiences crucial for their development. This issue is particularly detrimental to children with developmental delays, posing greater challenges for caregivers. These children often have fewer opportunities for therapy, education, and life participation, negatively affecting both the children's abilities and parental mental health. Research supports caregiver-centered interventions as beneficial for child development, reducing parent stress, and enhancing self-efficacy. However, there is a lack of multidisciplinary, relationship-enhancing programs for caregivers of children with developmental delays in early intervention clinical practice.

Purpose:This project aims to explore the effects of 'horticultural mediums', 'sensory experiences', and 'language guidance' on caregiver stress, self-efficacy, relationships, and parent-child conflict by involving both parents and children in gardening activities. Caregivers of children currently undergoing early intervention in outpatient clinics in the northern region will be recruited. Participants will be randomly assigned to either a gardening group (N=30) or a waiting group (N=30). The gardening group will engage in group gardening activities for six to eight weeks, while the waiting group will participate after an eight-week waiting period. Assessments before and after the intervention will include the Parental Competence Scale, Parenting Stress Index (Short Form), Pediatric Evaluation of Disability Inventory, and The Development of the Sensory Integration Functions Assessment Scale.

Data Analysis：The research data will be analyzed using SPSS (Version 20.0) with a significance level of 0.05. Results will be presented as mean ± standard deviation. Descriptive statistics will analyze basic data and assessment items of both groups. The Chi-square test will compare categorical data, while the Mann-Whitney U test and Kruskal-Wallis one-way ANOVA will compare outcomes within and between groups. Spearman's rank correlation will examine relationships between caregivers' and children's data, caregiver efficacy, stress, and children's sensory interaction.

ELIGIBILITY:
Inclusion Criteria:

* Children currently undergoing early intervention;
* Children experiencing sensory processing issues and caregivers (including grandparents and great-grandparents) seeking to establish parent-child relationships or enhance self-efficacy

Exclusion Criteria:

* Children don't accept early intervention.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-03-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Parenting Stress Index: Short form，PSI/SF | Change from Baseline at 6 weeks
  It designed for parents of children aged 0-12 years old in households experiencing parental stress, including parental distress, dysfunctional parent-child interaction, and difficult child behaviors. It consists of 36 items and has undergone factor analysis to establish content validity and construct validity. Each item on the scale demonstrates factor loadings greater than .30. The internal consistency of the entire scale ranges from .856 to .908 across its subscales, with a total scale reliability of .947, indicating high consistency in measuring the assessed content.
Parenting Sense of Confidence ，PSOC | Change from Baseline at 6 weeks
  This tool assesses parents' confidence and satisfaction in their role as caregivers, comprising 17 items rated on a 6-point Likert scale ranging from "1" (strongly agree) to "6" (strongly disagree), where higher scores indicate greater parental confidence. The scale demonstrates good internal consistency with an alpha coefficient of 0.82. It consists of two subscales: "Parenting Sense of Competence - Efficiency" (PSOC-E), which reflects feelings of frustration, anxiety, and motivation, and "Parenting Sense of Competence - Satisfaction" (PSOC-S), which assesses abilities, problem-solving skills, and satisfaction in the parental role.

SECONDARY OUTCOMES:
Chinese Version of Pediatric Evaluation of Disability Invertory | Change from Baseline at 6 weeks
  This tool is designed for functional assessment of children aged 6 months to 7 years and 6 months. It includes three different domains for evaluation. Given the study's focus on changes in children's participation and interaction abilities pre and post intervention, emphasis is placed on comparing the social functioning domain of the Functional Skills Assessment. Items assess abilities in communication, social interaction, household tasks, and community activities.
The Sensory Integration Functional Assessment Scale | Change from Baseline at 6 weeks
  It is designed for caregivers of children aged 3 to 10 years and 11 months. It assesses various aspects including postural and movement abilities, bilateral integration and sequencing of movements, sensory discrimination, sensory modulation, sensory seeking behaviors, attention and activity levels, and emotional/behavioral responses. The scale utilizes a five-point Likert scale and includes detailed items to evaluate children's performance across seven subscales.

CONTACTS AND LOCATIONS:
Overall Officials: ChiehYu Pan, Master, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No